CLINICAL TRIAL: NCT01637974
Title: Efficiency of INTERCOAT (Oxiplex/AP Gel) in Preventing Intrauterine Adhesion Formation in Hysteroscopic Surgery - a Prospective Double Blind Randomized Study
Brief Title: Efficiency of INTERCOAT (Oxiplex/AP Gel) in Preventing Intrauterine Adhesion Formation in Hysteroscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Moran Paz, M.D., Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CMC-11-0050-CTIL
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Asherman Syndrome; Endometrial Polyp; Uterine Myoma
MeSH Terms: conditions — Gynatresia; Myofibroma

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- with INTERCOAT (Experimental): injection of intercoat into the euterine cavity at the end of hysteroscopy
  Interventions: Drug: INTERCOAT administration
- without INTERCOAT (No Intervention): without INTERCOAT

INTERVENTIONS:
Drug: INTERCOAT administration — Applying INTERCOAT in the intrauterine cavity at the end of the hysteroscopic surgery
  Other Names: INTERCOAT
  Arms: with INTERCOAT

SUMMARY:
The study purpose is to examine the influence of INTERCOAT in prevention of intra-uterine adhesions formation after any hysteroscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years
* Must be able to understand, read and sign consent form

Exclusion Criteria:

* Signs of infection upon admission
* Ongoing pregnancy
* Carcinoma of the uterus or cervix
* Recurrent PID
* Women admitted for endometrial ablation
* Women that gave birth 6 weeks ago
* Women participating in another study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2012-12; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Presence of intra-uterine adhesions in a follow up diagnostic hysteroscopy | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Carmel Medical Center, Haifa, Haifa District, Israel